CLINICAL TRIAL: NCT06556888
Title: Observatory of Immunological Thrombopenic Purpura in the Brest Region: Descriptive and Comparative Cross-sectional Study
Brief Title: Observatory of Immunological Thrombopenic Purpura in the Brest Region
Acronym: OPTIMIST
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0089
Record Dates: First submitted 2020-11-19; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Database of patients with ITP, diagnosed, treated and followed in the Brest University Hospital.

DETAILED DESCRIPTION:
Creation of a global clinical and biological database for all patients diagnosed, treated and followed for ITP in the University Hospital of Brest.

UHB is the regional reference center (competence center) on hemorrhagic diseases.

Dr Pan-Petesch, who is responsible of the local competence center, is affiliated to the national sector of auto-immune cytopenias CERECAI-MARIH).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ITP agree to participate

Exclusion Criteria:

* Other thrombocythopenia other than ITP
* Patients Under guardianship
* Patients without national social security

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with ITP diagnosed, treated or followed at UHB
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2039-11-30 (Estimated)

PRIMARY OUTCOMES:
Description chronicity | 1 year
  Identification/description of risk factors of chronicity
Description treatment responses | 1 year
  Identification/ description of risk factors of bad responses

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Pan-Petesch, MD, Principal Investigator — UHB
Locations (1):
- Hematology Department - Institute of Oncology and Hematology, University Hospital of Brest, Brest, Brittany Region, France

IPD SHARING:
Plan to Share IPD: Undecided